CLINICAL TRIAL: NCT04827758
Title: Evaluation of a Screening Strategy for Sarcopenia: a Monocentric Prospective Cohort Study
Brief Title: Evaluation of a Screening Strategy for Sarcopenia: a Monocentric Prospective Cohort Study (STRAS)
Acronym: STRAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment to meet the objectives in time
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GHRMSA 1094; IDRCB 2020-A02364-35 (Other: French Health Organization)
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Sarcopenia
Keywords: sarcopenia; muscle strength; muscle mass; older people
MeSH Terms: conditions — Sarcopenia | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients hospitalized in the follow-up care and rehabilitation units (Other)
  Interventions: Procedure: Screening and diagnostic tests for sarcopenia

INTERVENTIONS:
Procedure: Screening and diagnostic tests for sarcopenia — All of the following tests and questionnaires will be performed :
  * SARC-F questionnaire,
  * measurement of muscle strengh by a grip test,
  * measurement of muscle mass by impedancemetry (ASM/size2),
  * 4-meter walking speed test,
  * Timed-Up and Go (TUG) test,
  * ADL (Activities of Daily Living) and IADL (Instrumental Activities of Daily Living) questionnaires.

SUMMARY:
The main objective of this study is to determine the prevalence of sarcopenia in patients hospitalized in the follow-up care and rehabilitation units of the geriatrics department of the Mulhouse French hospital.

DETAILED DESCRIPTION:
Secondary objectives

1. To assess the performance of the SARC-F questionnaire to screen for sarcopenia ;
2. To describe the characteristics of sarcopenic patients hospitalized in each follow-up care and rehabilitation unit (i.e. day hospital, full hospitalization);
3. To identify predictive factors of sarcopenia;
4. To determine, in the subgroup of patients hospitalized in the conventional follow-up care and rehabilitation unit (i.e. full hospitalization), the evolution of sarcopenia between admission and discharge of the following variables :

   1. muscle strength,
   2. muscle mass,
   3. functional ability,
   4. dependency.

Conduct of research

After receiving the written consent of the study participant, all of the following tests and questionnaires will be performed :

* SARC-F questionnaire,
* measurement of muscle strengh by a grip test,
* measurement of muscle mass by impedancemetry (ASM/size2),
* 4-meter walking speed test,
* Timed-Up and Go (TUG) test,
* ADL (Activities of Daily Living) and IADL (Instrumental Activities of Daily Living) questionnaires.

For patients in day hospital care, the study will end upon completion of these tests.

For patients hospitalized in the conventional follow-up care and rehabilitation unit (i.e. full hospitalization), a follow-up visit will be scheduled within 72 hours prior to the patient's discharge from the service, or at 3 months of hospitalization. The following tests and questionnaires will be performed during this visit:

* measurement of muscle strengh by a grip test,
* measurement of muscle mass by impedancemetry,
* 4-meter walking speed test,
* Timed Up and Go (TUG) test,
* ADL and IADL questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patient 60 years of age or older
* Patients hospitalized in the follow-up care and rehabilitation units (i.e. day hospital, full hospitalization) of the geriatrics department of the Mulhouse French hospital
* Patient who gave consent to participate in the study
* Affiliated or beneficiary of a social security scheme

Exclusion Criteria:

* Patient admitted for palliative care
* Bedridden patient
* Patient with major neurocognitive disorders preventing impedancemetry or grip test from being performed, or any other medical condition preventing impedancemtery or grip test from being performed
* Patient under legal protection
* Patient with an unstable psychiatric disorder
* Patient under guardianship or curatorship
* Patient already included in the study during a previous hospitalization

Secondary exclusion criteria :

- For patients hospitalized in the conventional follow-up care and rehabilitation unit (i.e. full hospitalization), impedancemtry or grip test not performed within 7 days of admission.

Patients excluded secondarily will not be replaced.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Number of patients with sarcopenia | Enrollment
  The diagnosis of sarcopenia will be established according to the 2018 criteria of the European Working Group On Sarcopenia in Older People (EWGSOP2) based on the evaluation of muscle strength and muscle mass. Sarcopenia will be defined by an abnormal value measured by a grip test and confirmed by an abnormal value of the ASM/size2 ratio measured by impedancemetry.

SECONDARY OUTCOMES:
Sensitivity, specificity, positive and negative predictive value of the SARC-F questionnaire | Enrollment
Characteristics of sarcopenic patients hospitalized in each follow-up care and rehabilitation unit (i.e. day hospital, full hospitalization) | Enrollment
Muscle strength | Hospital discharge assessed up to 3 months
  In the subgroup of patients hospitalized in the conventional follow-up care and rehabilitation unit (i.e. full hospitalization), the evolution of muscle strength between admission and discharge will be assessed by a grip test. For patients hospitalized for more than 3 months, the grip test will be performed at 3 months.
Muscle mass | Hospital discharge assessed up to 3 months
  In the subgroup of patients hospitalized in the conventional follow-up care and rehabilitation unit (i.e. full hospitalization), the evolution of muscle mass between admission and discharge will be assessed by the measurement of the ASM/size2 (impedancemetry) ratio. For patients hospitalized for more than 3 months, the measurement of muscle mass will be performed at 3 months.
4-meter walking speed test | Hospital discharge assessed up to 3 months
  In the subgroup of patients hospitalized in the conventional follow-up care and rehabilitation unit (i.e. full hospitalization), the evolution of the value of the 4-meter walking speed test between admission and discharge will be assessed. For patients hospitalized for more than 3 months, the 4-meter walking speed test will be performed at 3 months.
Timed-Up and Go test (TUG) | Hospital discharge assessed up to 3 months
  In the subgroup of patients hospitalized in the conventional follow-up care and rehabilitation unit (i.e. full hospitalization), the evolution of the value of the TUG test between admission and discharge will be assessed. For patients hospitalized for more than 3 months, the TUG test will be performed at 3 months.
ADL (Activities of Daily Living) questionnaire | Hospital discharge assessed up to 3 months
  In the subgroup of patients hospitalized in the conventional follow-up care and rehabilitation unit (i.e. full hospitalization), the ADL questionnaire will also be performed at hospital discharge, or at 3 months for patients hospitalized for more than 3 months.
IADL (Instrumental Activities of Daily Living) questionnaire | Hospital discharge assessed up to 3 months
  In the subgroup of patients hospitalized in the conventional follow-up care and rehabilitation unit (i.e. full hospitalization), the IADL questionnaire will also be performed at hospital discharge, or at 3 months for patients hospitalized for more than 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier SIRLIN, MD, Principal Investigator — Groupe Hospitalier de la Region de Mulhouse et Sud Alsace
Locations (1):
- GHRMSA - Hôpital Emile MULLER, Mulhouse, France